CLINICAL TRIAL: NCT02781948
Title: Evaluation of the Repeatability and Reproducibility of Corneal Epithelial Thickness Mapping With iVue SD-OCT
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-50997
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-05

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Not having any history of refractive surgery, contact lens, dry eye or pathology
  Interventions: Device: Optical Coherence Tomography
- Corneal condition: History of refractive surgery, contact lens, dry eye or keratoconus
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography

SUMMARY:
Evaluate the repeatability and reproducibility of iVue for measuring the total corneal thickness, the epithelial thickness, and the stromal thickness in normal subjects and patients with various corneal conditions.

ELIGIBILITY:
Inclusion Criteria:

Normal

* Able and willing to provide consent.
* Able and willing to complete required exams. Corneal conditions
* Able and willing to provide consent.
* Able and willing to complete required exams.
* History of refractive surgery, contact lens, dry eye or keratoconus.

Exclusion Criteria:

Normal

* History of refractive surgery, contact lens, dry eye or pathology.
* Blepharitis or meibomitis
* Unable to complete required exams. Corneal conditions
* Unable to complete required exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Epithelial thickness | Day 1

SECONDARY OUTCOMES:
Corneal thickness | Day 1

OTHER OUTCOMES:
Stromal thickness | Day 1